CLINICAL TRIAL: NCT03234140
Title: Constitutional Genetics to Predict Prognostic and Somatic Alterations in Follicular Lymphoma
Brief Title: Constitutional Genetics in Follicular Lymphoma
Acronym: CONPIL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0212
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Follicular Lymphoma; Genetic Predisposition to Disease
MeSH Terms: conditions — Lymphoma, Follicular; Genetic Predisposition to Disease | interventions — Genome-Wide Association Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group "Genome Wide Association Studies": Patients are adults, male or female, with a follicular lymphoma, homogeneously treated by immunochemotherapy included in one of the following cohorte :
  * PRIMA Cohort : phase III (Sponsor LYSARC, France; NCT00140582): N=396
  * RELEVANCE Cohort : phase III (Sponsor LYSARC, France; NCT01476787 ): N=441
  * FOLL05 Cohort: phase III (Sponsor Italian lymphoma Foundation, Italy; NCT00774826): N=229
  * MER1 Cohorts : prospective, observational (Sponsor Mayo Clinic, USA; IRB#09-001987): N=178
  * MER2 Cohorts : prospective, observational (Sponsor Mayo Clinic, USA; IRB#09-001987):N=321
  Using the Genome wide association studies (GWAS) approach on these 1,565 patients, the project plan to identify new prognostic markers. These markers will then be analyzed to decipher the impact of host genetics on somatic alterations and tumor biology, using public or matched patient data.
  Interventions: Genetic: Genome Wide Association Studies
- Group "EPIC": Patients are adults, male or female, included in the EPIC Cohort (European Prospective Investigation Into Cancer and Nutrition study between 1992 and 2000. (Sponsor IARC, Lyon, France).
  The investigators plan to analyze the influence of single-nucleotide polymorphisms on circulating t(14;18) levels in these 318 healthy individuals including 100 who will develop follicular lymphoma later on, and assess if these biomarkers are helpful to refine the identification of high-risk follicular lymphoma individuals.
  Interventions: Genetic: Single-nucleotide polymorphisms's genotyping

INTERVENTIONS:
Genetic: Genome Wide Association Studies — Using the Genome wide association studies (GWAS) approach on these 1,565 patients, the project plan to identify new prognostic markers. These markers will then be analyzed to decipher the impact of host genetics on somatic alterations and tumor biology, using public or matched patient data.
  Groups: Group "Genome Wide Association Studies"
Genetic: Single-nucleotide polymorphisms's genotyping — Analyze of the influence of single-nucleotide polymorphisms on circulating t(14;18) levels
  Groups: Group "EPIC"

SUMMARY:
Follicular lymphoma is the second most common adult B-cell lymphoma. The acquisition of the t(14;18) translocation is the genetic hallmark of Follicular lymphoma. However, 50% to 70% of healthy individuals harbor low levels of circulating t(14;18)-positive cells but will never develop Follicular lymphoma. It was observed that individuals who developed Follicular lymphoma showed a higher t(14;18) frequency than controls (Roulland et al., J Clin Oncol 2014). High t(14;18) frequency in blood from healthy individuals could be a predictive biomarker for Follicular lymphoma development. Genetic instability of those t(14;18)+ B-cells as well as failure of the micro-environment to control the proliferation of these cells are proposed mechanisms linking these lymphoma precursors to true lymphoma cells. The prognosis of Follicular lymphoma patients has been significantly improved mainly with the development of anti-CD20 monoclonal antibodies, with a current median overall survival over 15 years. However, this lymphoma remains an incurable disease. The most commonly used tool for prognostication of patients with Follicular lymphoma is the Follicular Lymphoma International Prognostic Index (FLIPI) based on conventional clinical and pathology parameters. Although it has clinical utility, the Follicular Lymphoma International Prognostic Index does not reflect the biologic heterogeneity of Follicular lymphoma. First-degree relatives of Follicular lymphoma had a fourfold increased risk of Follicular lymphoma suggesting a genetic etiology.

Using the Genome wide association studies (GWAS) approach on Follicular lymphoma cohorts of 1,565 patients, the project plan to identify new prognostic markers. These markers will then be analyzed to decipher the impact of host genetics on somatic alterations and tumor biology, using public or matched patient data. The investigators also plan to analyze the influence of single-nucleotide polymorphisms on circulating t(14;18) levels in 318 healthy individuals included in EPIC cohort that will develop Follicular lymphoma later on, and assess if these biomarkers are helpful to refine the identification of high-risk Follicular lymphoma individuals.

ELIGIBILITY:
Group "Genome Wide Association Studies"

Inclusion Criteria:

* Follicular lymphoma treated in first line therapy treated by immunochemotherapy (PRIMA, FOL05, MER1 and 2, control arm of RELEVANCE trial)
* Follicular lymphoma treated in first line therapy by Rituximab and Lenalidomide as part of the investigational arm of RELEVANCE trial
* Available constitutional DNA samples for GWAS analysis with an accurate consent form for such genetic study
* Available biological and clinical characteristics at diagnosis with a follow-up of the patient for event free survival analysis
* 18 years of age or older

Exclusion Criteria:

* A non-follicular lymphoma histology according to WHO 2016 classification (grade 1, 2, 3a follicular lymphoma)
* Relapsed follicular lymphoma
* Patients without an accurate consent form for constitutional genetic study
* Patients with no available biological or clinical data and follow-up for the outcome analysis

Group "EPIC"

Inclusion Criteria:

* Included in the EPIC Cohort (European Prospective Investigation into Cancer and nutrition study between 1992 and 2000)
* Available constitutional DNA samples with an accurate consent form for such genetic study
* 18 years of age or older

Exclusion Criteria:

* Patients without an accurate consent form for constitutional genetic study
* Patients with no available biological or clinical data and follow-up for the outcome analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group "Genome Wide Association Studies" :
  Patients are adults, male or female, with a follicular lymphoma, homogeneously treated by immunochemotherapy included in one of the following cohorte :
  * PRIMA Cohort : phase III (Sponsor LYSARC, France; NCT00140582): N=396
  * RELEVANCE Cohort : phase III (Sponsor LYSARC, France; NCT01476787 ): N=441
  * FOLL05 Cohort: phase III (Sponsor Italian lymphoma Foundation, Italy; NCT00774826): N=229
  * MER1 Cohorts : prospective, observational (Sponsor Mayo Clinic, USA; IRB#09-001987): N=178
  * MER2 Cohorts : prospective, observational (Sponsor Mayo Clinic, USA; IRB#09-001987):N=321
  Group "EPIC" :
  Patients are adults, male or female, included in the EPIC Cohort (European Prospective Investigation Into Cancer and Nutrition study between 1992 and 2000. (Sponsor IARC, Lyon, France).
Sampling Method: Probability Sample
Enrollment: 1883 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 1 year
  Event Free Survival for follicular lymphoma patients treated with modern immunochemotherapy in five cohorts is the primary end point defined as the time from the diagnosis or randomization to the date of progression, relapse, re-treatment, or death from any cause.
  Two steps analysis, with a discovery cohort and a validation cohort :
  The discovery cohorts that the investigators plan to study are a subset of patients with available deoxyribonucleic acid samples of two prospective phase III trials (PRIMA (NCT00140582) (N=396) and FOLL-05 (NCT00774826) (N=229), and one prospective observational cohort SPORE of the University of Iowa-Mayo Clinic (MER1; N=178). A GWAS will then be performed on a subset of patients with available deoxyribonucleic acid of two validation cohorts (Prospective observational SPORE MER2; N=321, phase III trial RELEVANCE, NCT01476787, N=441).

SECONDARY OUTCOMES:
Somatic alterations and tumor biology | 2 years
  In order to better decipher the impact of host genetics on somatic alterations and tumor biology and understand the physiological function of the single-nucleotide polymorphism identified from the primary outcome measure, we will study the link between the molecular profiles of the tumor and the prognostic single-nucleotide polymorphism. This will be performed on samples of the PRIMA and MER studies, for which we have access to somatic and constitutive data.
  In parallel, we will investigate the relation between known susceptibility single-nucleotide polymorphism and the level of the t(14 ;18) translocation. The latter analysis will be performed on EPIC samples (European Prospective Investigation Into Cancer and Nutrition), comparing healthy individuals to individuals who developed a follicular lymphoma. Finally, we will assess the effect of susceptibility single-nucleotide polymorphism on somatic molecular profiles on PRIMA and MAYO cohorts.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Hématologie Clinique, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No